CLINICAL TRIAL: NCT01300429
Title: Molecular Determinants of Acquired Clinical Resistance to Crizotinib in Non-small Cell Lung Cancer Harboring a Translocation or Inversion Event Involving the ALK Gene Locus
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-014
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer
Keywords: core biopsy; Resistance to Crizotinib; Non-small Cell Lung Cancer; 11-014
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue

GROUPS / COHORTS (1):
- patients with Non Small Cell Lung cancer: This is a protocol to obtain and/or analyze tissue specimens of patients with NSCLC harboring an activating ALK inversion or translocation that have had a previous clinical response to tyrosine kinase inhibitor therapy and subsequently experience progressive disease. The tissue will be used to identify changes in the ALK gene that are acquired during treatment with an ALK TKI and may account for acquired resistance.
  Interventions: Genetic: obtain tissue specimens

INTERVENTIONS:
Genetic: obtain tissue specimens — One core biopsy specimen will be placed in formalin and processed for cytogenetic and FISH analyses as well as DNA for ALK sequencing. The second core biopsy specimen will be immediately frozen in liquid nitrogen and stored in a -80 degree freezer for research specimen. Collection will be performed on-site at the time of the procedure.

SUMMARY:
The purpose of this study is to try to learn more about how small molecule kinase inhibitor medications work in treating lung cancer. Crizotinib (PF-02341066) is a drug that has been shown to shrink tumors in some patients with lung cancer. While the investigators know how this drug works to stop the growth of tumors that depend on change in the gene named ALK (also called EML4-ALK), the investigators do not know why the drug stops working. The investigators would like to examine the tumor to help us better understand why crizotinib has stopped working as well as it once did. The tumor will be examined with multiple tests to look for the reason that crizotinib stopped working.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histologically proven diagnosis of NSCLC at MSKCC Tumor positive for a translocation or inversion event involving the ALK gene locus
* Clinical response to treatment with crizotinib as defined by either:

Radiographic partial or complete response defined by RECIST or WHO

OR:

Radiographic stable disease for at least 8 weeks

* Radiographic progression of disease amenable to biopsy while on treatment with crizotinib as defined by RECIST or WHO
* Signed informed consent

Exclusion Criteria:

* Deemed by their treating physician to be medically unfit for biopsy
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen by the Thoracic Oncology Service who have been diagnosed with an ALK mutant NSCLC and treated with an ALK kinase inhibitor who have experienced objective regression by RECIST, WHO, or clinical criteria and who then progress will be screened for this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-02-08 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
the frequency of acquired mutations | 2 years
  ALK sequence from tumor tissue pre-treatment in patients that respond to crizotinib will be compared to ALK sequence in tumor tissue after the development of resistance when there is persistence of the original ALK inversion or translocation event.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2012-07-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT01300429/ICF_000.pdf